CLINICAL TRIAL: NCT06319482
Title: Evaluating and Comparing the Adherence of Proactive Management Therapy for Sleep Apnea
Brief Title: The Adherence of Proactive Sleep Apnea Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovaResp Technologies Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Adherence Study
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proactive CPAP Therapy (Intervention) (Experimental): Patients will undergo CPAP enabled with proactive therapy.
  Interventions: Device: Proactive CPAP Therapy
- Conventional APAP Therapy (Control) (Active Comparator): Patients will undergo conventional APAP therapy.
  Interventions: Device: Conventional APAP Therapy

INTERVENTIONS:
Device: Proactive CPAP Therapy — CPAP machine uses Artificial Intelligence to make predictions and preventions of future apneic events to auto-adjust pressure.
  Arms: Proactive CPAP Therapy (Intervention)
Device: Conventional APAP Therapy — CPAP machine relies on the detection of respiratory events to determine how to react and auto-adjust pressure.
  Arms: Conventional APAP Therapy (Control)

SUMMARY:
The goal of this clinical trial is to compare the adherence to Positive Airway Pressure (PAP) therapy for newly diagnosed Obstructive Sleep Apnea (OSA) patients. The main question(s) it aims to answer are:

1. To compare the adherence of proactive therapy and conventional Automatic-PAP (APAP) therapy short-term (3 months) and long-term (12 months) for newly diagnosed OSA patients.
2. To compare health outcomes (AHI, nightly usage, leak, and patient-reported outcomes) between proactive therapy and conventional APAP therapy.

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled superiority trial on newly diagnosed patients with obstructive sleep apnea. Each participant will be provided with a APAP device. The devices assigned to the test group will be modified to deliver the proactive therapy using Artificial Intelligence (AI). Devices assigned to the control group will deliver the conventional APAP therapy. A sleep technician will be in regular contact with participants and track the time spent interacting with each participant. At the conclusion of the first 3 months of the trial, participants who are acceptant to therapy will be asked if they would like to continue participating for an additional 9 months. Data will be collected by the PAP device and a series of self-reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Must have a new diagnosis of moderate or severe OSA (i.e., AHI > 15 events/hour).
* Must be 18-70 years old.
* No history of self-reported, uncontrolled, severe cardiovascular or neurological issues.
* Must be able to comply with all study requirements as outlined in the consent form.
* Must be able to follow the directions of the study doctor and research team.
* Must be able to understand English and be willing to provide informed consent.

Exclusion Criteria:

* Prior use of PAP machines.
* Subjects actively using bi-level PAP or require oxygen therapy.
* Subjects who are medically complicated or who are medically unstable ( i.e., cancer, dementia, unstable cardiac or respiratory disease, or unstable psychiatric illness).
* Potential sleep apnea complications that, in the opinion of the clinician, may affect the health and safety of the participant.
* Inability or unwillingness to given written informed consent.
* Neuromuscular disease, hypoglossal-nerve palsy, severe restrictive or obstructive pulmonary disease, moderate-to-severe pulmonary arterial hypertension, severe valvular heart disease, New York Heart Association class III or IV heart failure, recent myocardial infarction or severe cardiac arrhythmias (within the past 6 months), persistent uncontrolled hypertension despite medication use, active psychiatric disease, and coexisting non-respiratory sleep disorders that would confound functional sleep assessment.
* Pregnancy, planning to attempt to become pregnant, or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
Adherence | 3-12 months
  Calculated as at least 70% compliance (at least 4 hrs), in 30 days

SECONDARY OUTCOMES:
Apnea-Hypopnea Index | 3-12 months
  Calculated as the mean number of apnea and hypopnea events throughout the night in events/hr.
CPAP Therapy Usage | 3-12 months
  Calculated as the mean device usage by the patient throughout the night.
Self-assessed sleep outcomes | 3-12 months
  Patients will be requested to fill out a questionnaire to help evaluate their sleepiness before and after therapy.
  Scale: Epworth Sleepiness Scale on a 7-point scale, higher values meaning worse outcome.
Self-assessed functional outcomes | 3-12 months
  Patients will be requested to fill out a questionnaire to help evaluate their functional outcomes of sleep before and after therapy.
  Scale: Functional Outcomes of Sleep Questionnaire on a 7-point scale, higher values meaning better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- NovaResp Technologies Inc., Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No